CLINICAL TRIAL: NCT03047733
Title: Comparison of Cyclic On-off and Continuous Excimer Laser Treatment for Vitiligo: A Randomized Controlled Non-inferiority Trial
Brief Title: Comparison of Cyclic On-off and Continuous Excimer Laser Treatment for Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jae Min Sung, Resident of the department of dermatology, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AJIRB-MED-DE3-15-151
Record Dates: First submitted 2017-02-05; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Dermatologic Disease; Vitiligo
Keywords: Vitiligo; 308 nm excimer laser
MeSH Terms: conditions — Skin Diseases; Vitiligo | interventions — Tacrolimus; Ointments

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, split-body, non-inferiority trial.
  Patients with stable symmetric vitiligo were enrolled. The paired symmetric vitiliginous lesions were randomized to either the continuous or the cyclic on-off excimer laser treatment.
  Total duration of study was 9 months.
  In cyclic on-off excimer laser treatment, the cycle was arbitrarily determined that one cycle consists of a 2-month treatment period (on) and a consecutive 1-month intermission period (off).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- continuously excimer laser treatment (Active Comparator): In this group, lesions treated twice weekly through out the whole trial length (9 months).
  Application of topical tacrolimus 0.1% ointment through out the whole trial length (9 months).
  Interventions: Device: The XTRAC Excimer Laser System; Drug: Topical tacrolimus 0.1% ointment
- cyclic excimer laser treatment (Experimental): In this group, one cycle consists of a 2-month treatment period (on) and a consecutive 1-month intermission period (off).
  Total 3 cycles of cyclic treatment through out the whole trial length (9 months). During the treatment period, lesions treated twice weekly.
  Application of topical tacrolimus 0.1% ointment through out the whole trial length (9 months).
  Interventions: Device: The XTRAC Excimer Laser System; Drug: Topical tacrolimus 0.1% ointment

INTERVENTIONS:
Device: The XTRAC Excimer Laser System — Initial irradiation dose was 50 mJ/cm2 on face and 100 mJ/cm2 on trunk and extremities. If there had not been minimal asymptomatic erythema, energy level was escalated by 50 mJ/cm2.
  Other Names: XTRAC Velocity 400
Drug: Topical tacrolimus 0.1% ointment — Application of topical tacrolimus 0.1% ointment on the both lesions once daily.

SUMMARY:
OBJECTIVE: To investigate the efficacy of the cyclic on-off treatment compared to the conventional continuous excimer laser treatment.

DESIGN: A randomized, controlled, split-body, non-inferiority study. SETTING: The trial was performed in two tertiary health care centers in Korea.

PARTICIPANT: Twelve patients (16 pairs of lesions) with stable symmetric vitiligo less than 5 years' disease duration were enrolled.

INTERVENSION: The paired symmetric vitiliginous lesions were randomized to either the continuous or the cyclic on-off treatment. All lesions were treated twice weekly for 9-month: continuously, or cyclically with 2-month treatment and 1-month intermission (total 3 cycles). Topical tacrolimus was applied throughout the trial.

OUTCOME MEASURES: The repigmentation was assessed using an image analysis program with clinical photographs. The primary outcome was mean difference of repigmentation rates and the non-inferiority margin was set at 10%. During intermission period, the clinical changes such as loss of repigmentation or worsening of the vitiligo lesions were assessed.

DETAILED DESCRIPTION:
[Study design and population] A randomized, controlled, split-body, non-inferiority trial was designed.

After obtaining informed consent, 12 patients with stable symmetric vitiligo less than 5 years' disease duration were enrolled.

The patients taking systemic steroids or having enlarging lesions were excluded. The paired symmetric vitiliginous lesions were randomized to either the continuous or the cyclic excimer laser treatment.

Total duration of study was 9 months.

In cyclic excimer laser treatment, the cycle was arbitrarily determined that one cycle consists of a 2-month treatment period (on) and a consecutive 1-month intermission period (off) (total 3 cycles during the trial).

[Treatment protocol]

The lesions were treated twice a week. Initial irradiation dose was 50 mJ/cm2 on face and 100 mJ/cm2 on trunk and extremities. If there had not been minimal asymptomatic erythema, energy level was escalated by 50 mJ/cm2. In cyclic treatment, the treatment resumed after intermission with the previously used irradiation dose.

Topical tacrolimus 0.1% ointment was applied in both twice daily throughout whole length of the trial.

[Assessment and primary outcome] Photographic documentation of lesions was conducted every month and the degree of repigmentation was assessed with a repigmentation rate (%) from the baseline by using an image analysis program (Digital Researcher for Vitiligo Area Evaluation, Dr. VAE, Korea).

An intention-to-treat analysis was planned, and last observation carried forward method was applied to impute the missing value in the presence of dropouts.

The primary outcome was mean difference of quantitative changes in repigmented area between continuous and cyclic on-off treatment. The non-inferiority margin was set at 10%. During intermission period in the cyclic treatment, the clinical changes such as loss of repigmentation or worsening of the vitiligo lesions were assessed.

[Statistical analysis] All statistical analyses were conducted using R 3.2.4 (R Foundation for Statistical Computing, Austria) and a P value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symmetric vitiligo
* Patients with less than 5 years' disease duration

Exclusion Criteria:

* The patients taking systemic steroids
* The patients with currently enlarging lesions
* The patients who cannot follow the treatment schedule

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Mean difference of quantitative changes in repigmented area between continuous and cyclic on-off treatment. | Through study completion, an average of 9 months
  The degree of repigmentation was assessed with a repigmentation rate (%) with clinical photographs by using an image analysis program (Digital Researcher for Vitiligo Area Evaluation, Dr. VAE, Korea).

CONTACTS AND LOCATIONS:
Overall Officials: HEE YOUNG KANG, M.D., Ph.D., Study Director — Ajou University School of Medicine
Locations (1):
- Ajou university hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang XY, He YL, Dong J, Xu JZ, Wang J. Clinical efficacy of a 308 nm excimer laser in the treatment of vitiligo. Photodermatol Photoimmunol Photomed. 2010 Jun;26(3):138-42. doi: 10.1111/j.1600-0781.2010.00509.x. PMID 20584252
- [Background] Hofer A, Hassan AS, Legat FJ, Kerl H, Wolf P. Optimal weekly frequency of 308-nm excimer laser treatment in vitiligo patients. Br J Dermatol. 2005 May;152(5):981-5. doi: 10.1111/j.1365-2133.2004.06321.x. PMID 15888156
- [Background] Park KK, Liao W, Murase JE. A review of monochromatic excimer light in vitiligo. Br J Dermatol. 2012 Sep;167(3):468-78. doi: 10.1111/j.1365-2133.2012.11008.x. Epub 2012 Aug 8. PMID 22524428
- [Result] Aberdam E, Romero C, Ortonne JP. Repeated UVB irradiations do not have the same potential to promote stimulation of melanogenesis in cultured normal human melanocytes. J Cell Sci. 1993 Dec;106 ( Pt 4):1015-22. doi: 10.1242/jcs.106.4.1015. PMID 7907336